CLINICAL TRIAL: NCT02468544
Title: Development and Feasibility Testing of a Mobile Phone-Based HIV Primary Care Engagement Intervention
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left the institution prior to enrollment of the first participant.
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAO7902
Record Dates: First submitted 2015-05-31; First posted 2015-06-11 (Estimated); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: HIV; Adherence
Keywords: Engagement in care; mHealth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Intervention Study (Experimental): All participants will receive individualized text messages based on a schedule determined during the development and refinement of the mHealth text messaging intervention (i.e., once or twice a week). All participants will receive text messages for: 1) medication reminders, 2) appointment reminders, and 3) text messages addressing barriers (educational information to improve HIV knowledge) or promoting facilitators (e.g., routinizing taking of HIV antiretroviral medication) of care engagement. Each participant will complete baseline assessments, and will select their preferences for personalized messages on the day of baseline assessments. Text messages will be deployed for the duration of the 30-day trial. Participants will be followed-up at the completion of the 30-day intervention. Each participant will be asked to complete a follow-up survey, including questions on the acceptability of the mHealth intervention.
  Interventions: Other: Text messaging

INTERVENTIONS:
Other: Text messaging — Text messaging mHealth intervention to improve HIV Primary Care Engagement among clients of methadone maintenance treatment programs who are living with HIV.

SUMMARY:
This is an open-trial pilot study in which adult methadone maintenance treatment patients who are living with HIV but are not engaged in HIV primary care (i.e., missed appointments, non-adherence to medication) will be recruited to participate in a HIV primary care engagement study. The purpose of this study is to develop and test the feasibility and acceptability of a mobile phone-based health (mHealth) text messaging intervention to improve engagement in HIV primary care among substance abusing populations with HIV.

ELIGIBILITY:
Inclusion Criteria:

* Client of a methadone maintenance treatment program
* HIV positive (status confirmed by medical records)
* At least 18 years of age
* English speaking
* Comfortable using a mobile phone (to send and receive text messages)
* Lives in New York City
* Willingness to attend at least two design sessions
* Willingness to attend one usability testing session, and participate in a post-usability survey and exit interview.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03 (Estimated); Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Intervention | 30 days
  Acceptability of the intervention will be measured using the Technology Acceptance Model (TAM) scale.
Feasibility of Intervention | 30 days
  Feasibility of the intervention will be assessed focusing on study implementation, including recruitment and attrition rates.

SECONDARY OUTCOMES:
Efficacy of the intervention | 30 days
  Preliminary efficacy of the intervention will be measured using the HIV Treatment Adherence Self-Efficacy Scale (HIV-ASES) and the HIV appointment adherence questionnaire.

OTHER OUTCOMES:
Self-efficacy to self-manage HIV infection | 30 days
  Changes in self-efficacy to self-manage HIV infection will be measured using the self-management scale applied to persons with HIV/AIDS.
Improvements in HIV knowledge | 30 days
  Improvements in HIV knowledge will be measured by changes in HIV knowledge. We will use the HIV Knowledge Questionnaire (HIV-KQ-18) at baseline and at 30 days post baseline assessments to measure changes in HIV knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Jemima A. Frimpong, PhD., MPH, Principal Investigator — Columbia University
Locations (1):
- Acacia Network/Promesa, New York, New York, United States